CLINICAL TRIAL: NCT04252040
Title: A Randomized, Single Blind, Exploratory Study of the Acute Effects of Guided Imagery and Transcranial Direct Current Stimulation (tDCS) on Electroencephalogram (EEG) Alpha Brain Waves and Pain Levels in Women With Chronic Pelvic Pain
Brief Title: Open Label Extension Study of tDCS Plus Guided Imagery for Women With Chronic Pelvic Pain (CPP)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of participants. No enrollment
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Kenneth M Peters, MD, Director and Chair of the Department of Urology, Corewell Health East
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-382
Record Dates: First submitted 2020-01-27; First posted 2020-02-05 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Chronic Pelvic Pain
MeSH Terms: interventions — Imagery, Psychotherapy

STUDY DESIGN:
Intervention Model Description: This is an open label extension exploratory study. All eligible subjects will receive active tDCS with guided imagery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Active tDCS with guided imagery (Experimental): Subjects will receive 2 miliamps of electrical stimulation to the brain (transcranial direct stimulation-tDCS) for 20 minutes concurrently while listening to a guided imagery CD specifically designed for women with chronic pelvic pain.
  Interventions: Device: Active tDCS with guided imagery

INTERVENTIONS:
Device: Active tDCS with guided imagery — The subject will be positioned in the sitting/reclining position in a quiet room with lights dimmed. The tDCS device and audio headphones will be placed on the subject's head. The tDCS device to be used is the Soterix Medical 1X1 device using 2.0 mA of current. The electrodes that will be used will be standard sponge electrodes. The subject will listen to a scripted guided imagery CD specifically developed for women with chronic pelvic pain through the audio headphones. The guided imagery plus active tDCS arm will have 20 minutes of stimulation with 25 minutes of guided imagery.

SUMMARY:
This is an open label extension study trial of tDCS with a standardized guided imagery intervention. Up to 20 women with chronic pelvic pain, who completed participation in the initial randomized trial (IRB 2019-362) will be enrolled. Subjects will complete 5 tDCS treatments with guided imagery and a 1-week follow-up visit.

DETAILED DESCRIPTION:
Chronic pelvic pain (CPP) is a common and often debilitating in women. It occurs below the umbilicus and is severe enough to cause functional impairment or require treatment. Transcranial Direct Stimulation (tDCS) is a non-invasive brain stimulation technique. As tDCS modulates nerve activity and connectivity, it is also expected to cause measurable changes in brain activity. Guided imagery is a form of hypnosis using words to direct one's thoughts and attention to imagined sensations. Guided imagery has demonstrated efficacy in reducing pain related to many conditions including cancer pain, chronic lower back pain, and post-operative pain. More information is needed to evaluate the effects of tDCS and guided imagery in the treatment of chronic pelvic pain.

This study consists of one screening visit, 5 study intervention visits, and a 1-week follow-up visit. After obtaining informed consent, study staff will assess for changes in medical history an pelvic pain treatments since the end of participation in Part 1 (IRB 2019-362). Urine will be collected for urinalysis and a urine pregnancy test will be collected for women of childbearing potential. If urinalysis and pregnancy test are negative, subjects will complete questionnaires, vitals, and a baseline EEG will be conducted.

At the 5 interventional visits, transcranial direct stimulation (tDCS) with guided imagery will be delivered. A EEG will be completed after the 1st and 5th treatment visits. At each visit questionnaires will be administered and urine pregnancy test, if the woman is of childbearing potential. At the 1-week follow- up visit, an EEG will be performed, questionnaires administered.

ELIGIBILITY:
Inclusion Criteria:

* Study participants must have participated and completed: (IRB 2019-362) A Multi-Stage, Randomized, Single Blind, Pilot study of the Acute Effects of Guided Imagery and Transcranial Direct Current Stimulation (tDCS) on EEG Alpha Brain Waves and Pain Levels in Women with Chronic Pelvic Pain, referred to as Part
* Female
* Age 18 to 64 years
* Women must either be unable to become pregnant (are surgically sterile or postmenopausal) or must use an approved method of birth control throughout the study period.
* Self-reported CPP defined as pelvic pain that is non-cyclical and of at least 6 months duration and refractory to other treatments
* Subject agrees to not start any new treatment (medication or otherwise) throughout the treatment and follow up periods.
* Subject agrees to maintain stable doses of all current medications throughout the treatment and follow-up period.

Exclusion Criteria:

* History of seizures during the last 2 years or diagnosis of epilepsy
* Pacemaker
* Currently using tobacco
* Use of carbamazepine, oxcarbazepine, phenytoin, pramipexole or cabergoline within the past 6 months as self-reported
* Parkinson's Disease
* Any condition, including neurological or psychiatric illness, which per investigators' judgement may increase subject risk
* History of Hunner's lesions
* Lactation, pregnancy, or refusal to use medically approved/reliable birth control in women of child-bearing potential
* Sacral or pudendal Interstim® or spinal cord stimulator that is "on"
* Contraindications to tDCS stimulation (e.g. metal in the head, implanted brain medical devices, scalp wounds or infections, etc)
* History of head injury resulting in more than a momentary loss of consciousness during the last 2 years

Deferral Criteria

1. If a subject has a confirmed UTI per investigator's clinical judgment, she will be deferred until treatment is completed and symptoms resolve
2. Participating in another intervention study, or received an investigational drug or device within 4 weeks prior to screening
3. Subject received bladder hydrodistention within the past 12 weeks
4. Within the past four weeks, initiation of any new medications or any intravesical treatment for treatment of IC/BPS.
5. Within the past 24 weeks received any surgery or procedure which may impact the pelvic floor

   * Note: For the sake of preserving scientific integrity, one of more of the eligibility criteria have been left off this list posting while the trial is ongoing. A full list of eligibility criteria will be posted upon completion of the trial.

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03 (Estimated); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-17 (Actual)

PRIMARY OUTCOMES:
To assess changes in EEG alpha brain waves in women with CPP after 5 sessions of transcranial direct simulation (tDCS) administered concurrently with guided imagery (GI). | At 1-week follow up visit.
  Change in alpha wave frequency on EEG between baseline and after the 5th interventional treatment of tDCS with guided imagery.

SECONDARY OUTCOMES:
To assess changes in pain in women with CPP after 5 sessions of transcranial direct simulation (tDCS) administered concurrently with guided imagery (GI). | At 1-week follow-up.
  A 10-point VAS for pain will be utilized at screening to determine eligibility, and pre- and post-treatment to measure the short-term effects of each treatment. VAS is scored from 0-10.
To assess changes in urinary symptoms in women with CPP after 5 sessions of transcranial direct simulation (tDCS) administered concurrently with guided imagery (GI) as measured by the Overactive Bladder Questionnaire short form (OAB-q SF). | At 1-week follow-up visit.
  Changes in subject-reported bother related to overactive bladder symptoms as measured by the Overactive Bladder Questionnaire short form (OAB-q SF). The OAB-q SF consists of two scales assessing symptom bother and health-related quality of life (HRQOL) in patients with OAB. Each question is rated on a 6-point scale with 1 = not at all and 6= a very great deal.
To assess changes in urinary symptoms in women with CPP after 5 sessions of transcranial direct simulation (tDCS) administered concurrently with guided imagery (GI) as measured by the Interstitial Cystitis Symptom Index and Problem Index ICSI-PI). | At 1-week follow-up visit.
  The IC symptom and problem index measure urinary and pain symptoms and assess how problematic symptoms are for patients with IC/BPS. Scored (0-36). A higher score indicates greater severity of symptoms.
To assess changes in QOL in women with CPP after 5 sessions of transcranial direct simulation (tDCS) administered concurrently with guided imagery (GI). | At 1-week follow-up visit.
  The Global Response Assessments (GRA) for Pain and QOL will administered. GRA evaluates the subject's perceptions of overall improvement in symptoms on a 7-point scale (markedly worse, moderately worse, mildly worse, same, slightly improved, moderately improved, or markedly improved).

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth M Peters, MD, Principal Investigator — Beaumont Health
Locations (2):
- United States (2):
  - Beaumont Health System, Royal Oak, Michigan
  - Beaumont Hospital-Royal Oak, Royal Oak, Michigan

IPD SHARING:
Plan to Share IPD: No